CLINICAL TRIAL: NCT02463994
Title: A Pilot Study of MPDL3280A (PD-L1) Antibody Therapy and Hypofractionated Image-guided Radiotherapy (HIGRT) in Patients With Metastatic Non-Small Cell Lung Cancer
Brief Title: A Pilot Study of MPDL3280A and HIGRT in Metastatic NSCLC
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2015.005; HUM00100387 (Other: IRBMED)
Record Dates: First submitted 2015-05-29; First posted 2015-06-08 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MPDL3280A + HIGRT (Experimental)
  Interventions: Drug: MPDL3280A; Radiation: Hypofractionated Radiotherapy

INTERVENTIONS:
Drug: MPDL3280A — Patients will receive 1,200 mg I.V. Q 3 weeks of MPDL3280A until progression.
Radiation: Hypofractionated Radiotherapy — Hypofractionated Image-Guided Radiotherapy (HIGRT)

SUMMARY:
The purpose of this study is to find out whether a brief course of radiation therapy given to one area affected by the cancer will improve the chances of responding to immuno-therapy in the form of a medicine called MPDL3280A, an antibody against PD-L1. PD-L1 is expressed on lung cancers and is known to block the effects of the body's immune system in attacking the cancer. Blocking this PD-L1 has been shown to improve the body's immune cells to attack and kill the cancer cells in non-small cell lung cancer. The goal of this study is to see if prior treatment with radiation will allow improved recognition of the cancer by the body's immune cells in the presence of MPDL3280A.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form (ICF)
* Ability and willingness to comply with the requirements of the study protocol
* Age ≥18 years old
* ECOG (Eastern Cooperative Oncology Group) performance status (PS) of 0 or 1 (scores run from 0 to 5 where 0 denotes perfect health and 5 death).
* Patients with ECOG PS of 2, secondary to the underlying disease, may be enrolled.
* Patients with Stage IIIB (not eligible for definitive chemo-radiotherapy), Stage IV, or recurrent non-small cell lung cancer (NSCLC); patients with Stage IV NSCLC should have previously received platinum based doublet chemotherapy. Patients with a new diagnosis of Stage IV NSCLC are eligible if they have an initial requirement for palliative XRT for symptomatic lesion (example: painful bone lesion or obstructive airway).
* Patients must be candidates for palliative radiation.
* Measurable disease per mRECIST v1.1 Patients must have at least 1 distinct site of measurable disease, ≥ 1 cm in its largest diameter, in addition to the site that is being irradiated.
* Patients may have additional measurable and/or non-measurable but radiographically visible metastatic lesions (e.g. bone metastases).
* Patients with treated brain metastasis as long as neurologically stable and not on steroids for at least 12 weeks (see Exclusion criteria below for details).
* Patients must be candidates for PD-L1 Ab as determined by the treating physician
* At least 3 weeks must have elapsed from any prior chemotherapy, and the patient must have recovered from side effects to ≤ grade 1 toxicities.
* Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to the first study treatment (Cycle 1, Day 1):
* ANC (Absolute Neutrophil Count) ≥ 1500 cells/µL
* WBC (White Blood Cell) counts > 2500/µL
* Lymphocyte count ≥ 500/µL
* Platelet count ≥ 100,000/µL; for patients with hematologic malignancies, platelet count ≥ 75,000/µL
* Hemoglobin ≥ 9.0 g/dL
* Total bilirubin ≤ 1.5 x ULN with the following exception:
* Patients with known Gilbert disease who have serum bilirubin level ≤ 3 x ULN may be enrolled.
* AST (Aspartate Aminotransferase) and ALT (Alanine Aminotransferase) ≤ 3.0 x ULN with the following exception: Patients with liver involvement: AST and/or ALT ≤ 5 x ULN
* Alkaline phosphatase ≤ 2.5 x ULN with the following exception: Patients with documented liver involvement or bone metastases: alkaline phosphatase ≤ 5 x ULN
* Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min on the basis of the Cockcroft-Gault glomerular filtration rate estimation: (140 - age) x (weight in kg) x (0.85 if female) 72 x (serum creatinine in mg/dL)
* INR (International Normalized Ratio) and aPTT ≤1.5 x ULN
* This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation (such as low molecular weight heparin or warfarin) should be on a stable dose.
* For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use highly effective form(s) of contraception (i.e., one that results in a low failure rate [<1% per year] when used consistently and correctly) and to continue its use for 6 months after the last dose of MPDL3280A
* Representative tumor specimens in paraffin blocks (preferred) or at least 15 unstained slides, with an associated pathology report, requested at any time prior to study entry. Only tissue from core needle, punch, or excisional biopsy sample collection will be accepted. Fine-needle aspiration, brushing, and lavage samples are not acceptable. For all biopsy types, submitted blocks should have sufficient tissue to generate at least 15 sections, and tissue for which the pathology report specifies that the overall tumor content is low (e.g., "sparse" or "scant") is not acceptable. Tissue from separate time points (such as time of initial diagnosis and time of metastatic diagnosis) or from the multiple metastatic tumors may also be collected for a given patient, on the basis of availability.
* If archival tissue is either insufficient or unavailable, the patient may still be eligible if the patient can provide at least five unstained, serial slides or is willing to consent to and undergo a pre-treatment core or excisional biopsy sample collection of the tumor. Fine-needle aspiration, brushing, and lavage samples are not acceptable.

Exclusion Criteria:

* Any approved anticancer therapy, including chemotherapy, hormonal therapy, or radiotherapy, within 3 weeks prior to initiation of study treatment; however, the following are allowed:
* Hormone-replacement therapy or oral contraceptives.
* Herbal therapy > 1 week prior to Cycle 1, Day 1 (herbal therapy intended as anticancer therapy must be discontinued at least 1 week prior to Cycle 1, Day 1).
* Palliative radiotherapy for bone metastases < 2 weeks prior to Cycle 1, Day 1
* AEs from prior anticancer therapy that have not resolved to Grade ≤ 1 except for alopecia.
* Bisphosphonate therapy for symptomatic hypercalcemia.
* Use of bisphosphonate therapy for other reasons (e.g., bone metastasis or osteoporosis) is allowed.
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, cirrhosis, fatty liver, and inherited liver disease.
* Patients with acute leukemias, accelerated/blast-phase chronic myelogenous leukemia, chronic lymphocytic leukemia (except Rai-stage I), Burkitt lymphoma, plasma cell leukemia, or non-secretory myeloma
* Known primary CNS (Central Nervous System) malignancy or symptomatic CNS metastases
* Patients with asymptomatic untreated CNS disease may be enrolled after consultation, provided all of the following criteria are met:
* Evaluable or measurable disease outside the CNS
* No metastases to brain stem, midbrain, pons, medulla, cerebellum, or within 10 mm of the optic apparatus (optic nerves and chiasm)
* No history of intracranial hemorrhage or spinal cord hemorrhage
* No ongoing requirement for dexamethasone for CNS disease; patients on a stable dose of anticonvulsants are permitted
* No neurosurgical resection or brain biopsy within 28 days prior to Cycle 1, Day 1
* Patients with asymptomatic treated CNS metastases may be enrolled after consultation, provided all the criteria listed above are met as well as the following:
* Radiographic demonstration of improvement upon the completion of CNS-directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study
* No stereotactic radiation or whole-brain radiation within 28 days prior to Cycle 1, Day 1
* Screening CNS radiographic study ≥ 4 weeks from completion of radiotherapy and ≥ 2 weeks from discontinuation of corticosteroids
* Pregnancy, lactation, or breastfeeding
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Inability to comply with study and follow-up procedures
* History or risk of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis
* Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.
* Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible.
* Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:
* Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
* Rash must cover less than 10% of body surface area (BSA)
* Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%)
* No acute exacerbations of underlying condition within the last 12 months (not requiring PUVA [Psoralen Plus Ultraviolet A Radiation], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high potency or oral steroids)
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest CT scan
* History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* History of HIV infection or active hepatitis B (chronic or acute) or hepatitis C infection
* Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [Antibody to Hepatitis B Core Antigen] antibody test) are eligible.
* Patients positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* Active tuberculosis
* Severe infections within 4 weeks prior to Cycle 1, Day 1 including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection within 2 weeks prior to Cycle 1, Day 1
* Received oral or IV antibiotics within 2 weeks prior to Cycle 1, Day 1
* Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible.
* Major surgical procedure within 28 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure during the course of the study
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1 or anticipation that such a live attenuated vaccine will be required during the study
* Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine (e.g., FluMist) within 4 weeks prior to Cycle 1, Day 1 or at any time during the study.
* Malignancies other than disease under study within 5 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death and with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, or ductal carcinoma in situ treated surgically with curative intent) or undergoing active surveillance per standard-of-care management (e.g., CLL Rai Stage 0, prostate cancer with Gleason score ≤ 6, and PSA ≤10 mg/mL, etc.)

Medication-Related Exclusion Criteria:

* Prior treatment with anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway targeting agents
* Patients who have received prior treatment with anti-CTLA-4 may be enrolled, provided the following requirements are met:
* Minimum of 12 weeks from the first dose of anti-CTLA-4 and > 6 weeks from the last dose
* No history of severe immune-related adverse effects from anti-CTLA-4 (CTCAE Grade 3 and 4)
* Treatment with systemic immunostimulatory agents (including but not limited to IFN, IL-2) within 6 weeks or five half-lives of the drug (whichever is shorter) prior to Cycle 1, Day 1
* Treatment with investigational agent within 4 weeks prior to Cycle 1, Day 1 (or within five half-lives of the investigational product, whichever is longer)
* Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents) within 2 weeks prior to Cycle 1, Day 1
* Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled.
* The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation

Specific Exclusion Criteria:

* Patients having no distinct measurable lesions outside of the field of radiation.
* Previous radiotherapy to the lesion(s) of interest.
* Concurrent treatment with any other anti-neoplastic drug or concurrent participation in another therapeutic clinical trial
* Patients with EGFR/ALK/ROS-1+ lung adenocarcinoma.
* Uncontrolled tumor-related pain.
* Uncontrolled hypercalcemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
The number of participants that respond to a combination of HIGRT and MPDL3280A (PD-L1) | 5 years
  The primary outcome is overall response rate (ORR) to combination of HIGRT and MPDL3280A. The number of participants that respond to treatment will be determined. Response will be assessed by Response Evaluation Criteria in Solid Tumors (mRECIST) version 1.1, using primarily CT scans, immune response criteria and/or clinical benefit as assessed by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Nithya Ramnath, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (2):
- United States (2):
  - The University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Washington, Seattle, Seattle, Washington